CLINICAL TRIAL: NCT04865354
Title: Clinical Comparison of Two Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLE383-P005
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Results first posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Refractive Errors
Keywords: Contact Lenses; Disposable
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PRECISION1, then Clariti 1-Day (Other): Verofilcon A contact lenses worn first, with somofilcon A contact lenses worn second, as randomized. Each study lens type will be worn bilaterally (in both eyes) for 8 days in a daily disposable modality.
  Interventions: Device: Verofilcon A contact lenses; Device: Somofilcon A contact lenses
- Clariti 1-Day, then PRECISION1 (Other): Somofilcon A contact lenses worn first, with verofilcon A contact lenses worn second, as randomized. Each study lens type will be worn bilaterally (in both eyes) for 8 days in a daily disposable modality.
  Interventions: Device: Verofilcon A contact lenses; Device: Somofilcon A contact lenses

INTERVENTIONS:
Device: Verofilcon A contact lenses — Spherical soft contact lenses for daily disposable wear
  Other Names: PRECISION1
Device: Somofilcon A contact lenses — Spherical soft contact lenses for daily disposable wear
  Other Names: Clariti 1-Day

SUMMARY:
The purpose of this study is to compare the clinical performance of PRECISION1™ contact lenses to Clariti® 1 day contact lenses.

DETAILED DESCRIPTION:
Subjects will be expected to attend 3 study visits and wear the study lenses daily for at least 10 hours per day. On the day prior to Visits 2 and 3, subjects will be expected to wear the study lenses for at least 16 hours. The total duration of subject participation will be up to 22 days.

ELIGIBILITY:
Key Inclusion Criteria

* Successful wearer of spherical soft contact lenses with at least 3 months wearing experience, with a minimum wearing time of 5 days per week and 10 hours per day.
* Possess spectacles and willing to wear habitual spectacles for vision correction when study lenses are not worn, as needed.
* Willing to wear contact lenses for at least 16 hours on one of the days (day prior to each week 1 visit).
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Habitual PRECISION1, Clariti 1-Day, and DAILIES TOTAL1 contact lens wearers.
* Any monovision and multifocal lens wearers.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-06-27 (Actual); Study Completion 2021-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CDMA Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (8):
- United States (8):
  - Alcon Investigator 8106, San Francisco, California
  - Alcon Investigator 6565, Maitland, Florida
  - Alcon Investigator 6418, Tallahassee, Florida
  - Alcon Investigator 6614, Franklin Park, Illinois
  - Alcon Investigator 6645, Shawnee Mission, Kansas
  - Alcon Investigator 6402, Medina, Minnesota
  - Alcon Investigator 8046, Granville, Ohio
  - Alcon Investigator 8028, Wichita Falls, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 8 investigative sites in the United States.
Pre-assignment Details: Of the 170 enrolled, 3 subjects were exited prior to randomization as screen failures. This reporting group includes all randomized subjects (167).
Groups:
- PRECISION1, Then Clariti 1-Day: Verofilcon A contact lenses worn first, with somofilcon A contact lenses worn second, as randomized. Each study lens type was worn bilaterally (in both eyes) for 8 days in a daily disposable modality.
- Clariti 1-Day, Then PRECISION1: Somofilcon A contact lenses worn first, with verofilcon A contact lenses worn second, as randomized. Each study lens type was worn bilaterally (in both eyes) for 8 days in a daily disposable modality.
Period: First Wear Period (8 Days)
Arm/Group | PRECISION1, Then Clariti 1-Day | Clariti 1-Day, Then PRECISION1
Started | 83 | 84
Completed | 82 | 83
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Period: Second Wear Period (8 Days)
Arm/Group | PRECISION1, Then Clariti 1-Day | Clariti 1-Day, Then PRECISION1
Started | 82 | 83
Completed | 81 | 83
Not Completed | 1 | 0
Not completed — Protocol deviation, dispensed wrong powers | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All randomized subjects who are exposed to any study lenses evaluated in this study
Groups:
- Total: Total of all reporting groups
Arm/Group | PRECISION1, Then Clariti 1-Day | Clariti 1-Day, Then PRECISION1 | Total
Number analyzed (Participants) | 83 | 84 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (8.9) | 31.4 (7.5) | 31.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 62 | 116
  Male | 29 | 22 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 13
  Not Hispanic or Latino | 78 | 76 | 154
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 69 | 67 | 136
  Black or African American | 1 | 3 | 4
  Asian | 12 | 13 | 25
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 83 | 84 | 167

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Distance VA (logMAR) With Study Lenses
Description: Distance visual acuity (VA) was assessed with study lenses in place. VA was collected for each eye separately using logarithmic of the Minimum Angle of Resolution (logMAR) charts. A logMAR acuity of 0.0 corresponds to 20/20 Snellen acuity (normal visual acuity), with a negative value denoting better than 20/20 visual acuity.
Time Frame: Day 8, each study lens type
Population: Full Analysis Set: All randomized subjects who are exposed to any study lenses evaluated in this study with non-missing response (eye)
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Groups:
- PRECISION1: Verofilcon A contact lenses worn bilaterally (in both eyes) during Period 1 or Period 2, as randomized, for 8 days in a daily disposable modality
- Clariti 1-Day: Somofilcon A contact lenses worn bilaterally (in both eyes) during Period 1 or Period 2, as randomized, for 8 days in a daily disposable modality
Arm/Group | PRECISION1 | Clariti 1-Day
Number analyzed (Participants) | 164 | 164
Number analyzed (eyes) | 328 | 328
logMAR | -0.119 (0.0055) | -0.122 (0.0055)
Statistical Analysis 1: Comparison: PRECISION1 vs Clariti 1-Day; Test type: Non-Inferiority — Noninferiority to be concluded if least squares means difference upper confidence limit is less than 0.05; Since a noninferiority hypothesis is being tested, a p-value is not applicable. Confidence limit is being reported and compared to the noninferiority margin; LSM results based on general linear mixed effects model with terms for lens, period and sequence as fixed effects, subject as a random effect; Least Squares Mean Difference = 0.003, 95% CI 1-sided [upper limit 0.009], Standard Error of Mean 0.0034 — Difference = PRECISION1 minus Clariti 1-Day

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, up to 22 days.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of participants. This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study. Note: One subject (2 eyes) wore PRECISION1 in both periods and did not wear Clariti 1-Day.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses
- PRECISION1 Ocular; PRECISION1 Systemic: Events reported in this group occurred while exposed to the verofilcon A contact lenses
- Clariti 1-Day Ocular; Clariti 1-Day Systemic: Events reported in this group occurred while exposed to the somofilcon A contact lenses
Arm/Group | Pretreatment | PRECISION1 Ocular | PRECISION1 Systemic | Clariti 1-Day Ocular | Clariti 1-Day Systemic
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/334 | 0/167 | 0/332 | 0/166
Serious Adverse Events (participants affected / at risk) | 0/167 | 0/334 | 0/167 | 0/332 | 0/166
Other Adverse Events (participants affected / at risk) | 0/167 | 0/334 | 0/167 | 0/332 | 0/166

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2021-04-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT04865354/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/54/NCT04865354/SAP_001.pdf